CLINICAL TRIAL: NCT06875297
Title: A Comprehensive Cancer Genome Profiling to Detect Actionable Alteration Representative of Progression of Non-metastatic Prostate Cancer.
Brief Title: A Single-center Prospective Interventional Study on FPG500 in Non-metastatic Prostate Cancer Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IDTBD
Record Dates: First submitted 2025-03-04; First posted 2025-03-13 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a single-center prospective interventional study involving patients with histologically confirmed low-risk, high-risk and locally advanced PCa.
  Patients' treatment will be prompted according to international Guidelines and Good Clinical Practice. A cancer genome profiling with FPG 500 will be performed within these cohorts.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FPG500 test (Experimental): This is a single-center prospective interventional study involving patients with histologically confirmed low-risk, high-risk and locally advanced PCa.
  A cancer genome profiling with FPG 500 will be performed within these cohorts. Samples will be available from surgery for high-risk and locally advanced PCa, from prostate biopsy for low risk patients.
  Interventions: Diagnostic Test: FPG500

INTERVENTIONS:
Diagnostic Test: FPG500 — A cancer genome profiling with FPG500 will be performed on samples available from surgery or biopsy. Specimen are reviewed to assess tumor cell fraction. All H&E slides are digitized before nucleic acid extraction. Semi-automated process is used for DNA/RNA extraction, DNA fragmentation, quantification, library preparation, and sequencing. Profiling is done with the TruSight Oncology 500 assay, analyzing 523 genes for single nucleotide variants, insertions/deletions, copy number variations, and fusions/splicing variants in 55 genes. It also evaluates genomic signatures like microsatellite instability and tumor mutational burden. Sequencing data are processed using Illumina software and a custom pipeline. Post-sequencing quality control is performed. Variants are classified according to the Human Genome Variation Society and clinical actionability guidelines. Genomic report is reviewed by an institutional Molecular Tumor Board.

SUMMARY:
The search for clinically actionable alterations within the non-metastatic prostate cancer setting has been an overlooked issue so far. Genomic alterations predicting tumor progression or representative of micrometastatic spread could be crucial to prompt the correct treatment strategy, sequencing and possible intensification in the high-risk and locally advanced settings. Similarly, the definition of the genomic landscape in low-risk patients progressing to more aggressive disease could be of importance to prompt an immediate active treatment to those patients otherwise eligible to active surveillance.

A CGP program has been launched by the Fondazione Policlinico Universitario Agostino Gemelli IRCCS (FPG), a leading Italian research hospital (ID: FPG500, ethical approval number 3837) and it convers 10 cancer types. This program offers genomic testing of over 500 genes through an efficient in-house process. To now, a CGP from FPG 500 has been applied to cholangiocarcinoma, endometrial cancer, non-small cell lung cancer.

Investigators propose a prospective interventional single center study whose aim is to implement a comprehensive genome profiling (CGP) through this next generation sequencing (NGS) program for non-metastatic PCa and to define actionable mutations that correlate with tumor progression. The actionability relies on the opportunity to intensify treatment in non metastatic cases at risk of progression or to identify distant spread before it becomes biochemically and/or radiographically evident for high risk non metastatic cancers.

From previous research, a genomic profiling may reveal distinct mutations or gene expression patterns linked to metastasis, biochemical recurrence, and PSA persistence. Some of these genomics alterations may be associated with poorer outcomes in high-risk and locally advanced patients. Conversely, patients under active surveillance might exhibit a more stable genomic profile, with fewer mutations representative of aggressive disease. Expected outcomes will include the development of accurate prognostic tools, allowing for better-tailored treatment plans and early intervention strategies to manage disease progression.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven diagnosis of low-risk, or high-risk or locally advanced prostate cancer
* high-risk and locally advanced prostate cancer undergoing surgery
* low-risk prostate cancer undergoing active surveillance or surgery

Exclusion Criteria:

* previous or concomitant malignancies
* patients already undergoing androgen suppression or other medical treatments for prostate cancer

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2025-08-05 (Estimated); Primary Completion 2027-10-08 (Estimated); Study Completion 2029-08-07 (Estimated)

PRIMARY OUTCOMES:
Rate of patients with FPG500 mutations (ie AMP-ASCO-CAP Tier I-II) associated with biochemical relapse or PSA persistence after surgery | 3 years
  A raise in the PSA level is the first sign of disease progression for the whole non-metastatic PCa setting. After radical prostatectomy in high-risk patients, biochemical relapse anticipates radiographic progression and is a crucial point invoking re-staging and treatment decision making. A PSA doubling time below 8-10 months is significantly related to metastatic development and prostate cancer specific death (Smith MR, J Clin Oncol 2013;31:3800-3806).
  The primary endpoint is to identify actionable mutations related to BCR (or persisting PSA) after surgery for high-risk and locally advanced PCa.
Rate of patients with FPG500 mutations (ie AMP-ASCO-CAP Tier I-II) associated with cancer progression in low-risk pts undergoing active surveillance | 5 years
  The primary endpoint is to identify actionable mutations related to progression of low-risk PCa. From the study from Hamdy et al, the occurrence of clinical progression requiring active treatment is as high as 25% at 15 years.
  PCa cases with diagnosis of low-risk will be considered for FPG 500 genomic profiling from prostate biopsy to define mutations related to:
  - Upstage and/or upgrade of cancer during surveillance protocol

SECONDARY OUTCOMES:
Rate of patients with FPG500 mutations in high risk non-met pts - non-met definition based on conventional and/or PSMA/PET imaging - with fast radiographic progression after surgery, suggesting a micrometastatic status at diagnosis | 3 years
  Radiographic progression of cancers may relate with the development of symptoms and with an increased burden of cure to control clinical progression. FPG500 mutations relevant to this endpoint may suggest treatment anticipation /intensification after surgery or may be actionable of target treatment

CONTACTS AND LOCATIONS:
Overall Officials: maria chiara, Principal Investigator — Fondazione
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, UOC Urologia, Roma, Italy

REFERENCES:
- [Derived] Sighinolfi MC, Pallotta G, Assumma S, Panio E, Pinto F, Gavi F, Totaro A, Presutti S, Pasciuto T, Nero C, Del Re M, Tagliaferri L, Ciccarese C, Iacovelli R, Gabarrini A, Patel E, Moschovas MC, Patel V, Rocco B. A novel comprehensive cancer genome profiling for non-metastatic prostate cancer: study protocol with FPG500 to detect actionable alterations representative of progressive disease. BJU Int. 2025 Dec;136(6):1022-1027. doi: 10.1111/bju.70019. Epub 2025 Oct 10. PMID 41070807